CLINICAL TRIAL: NCT00822601
Title: A Controlled Study of rTMS Over Supplementary Motor Area (SMA) in Obsessive Compulsive Disorder
Brief Title: Study of Repetitive Transcranial Magnetic Stimulation Efficacy on Obsessive Compulsive Disorder (OCD)
Acronym: TMS-TOC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AOR07067
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2009-01

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Repetitive Transcranial Magnetic Stimulation; Supplementary Motor Area; Obsessive-Compulsive Disorder; Sham rTMS; Placebo-controlled; Randomized; Double-blind; fMRI; DSM-IV Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Device: rTMS
- 2 (Placebo Comparator)
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: rTMS — Arm 1 (experimental) : rTMS, 4 weeks of stimulation with RMT frequency 1Hz, intensity 100% of RMT for 20 minutes (1500 pulses), 5 minutes of trains with 2 minutes of intra-train intervals to both SMA. Treatment will be given 5 times a week for 4 weeks.
  Arms: 1
Device: Sham Comparator — sham rTMS (using a placebo coil), 4 weeks of stimulation, will mimic the active treatment mentioned above.
  Arms: 2

SUMMARY:
Our study's purpose is to show the efficacy of the transcranial magnetic stimulation (a non invasive method of cerebral modulation) in patients suffering from chronic obsessive compulsive disorder (OCD). This new method will be applied in 20 patients during 4 weeks (5 sessions each week), and its effects on OCD symptoms will be compared to those of a "sham" (=placebo) stimulation applied with the same process in 20 other patients, randomly assigned to the comparison group. The maintenance of the therapeutic effects will be explored during 8 weeks following the end of the treatment. In addition to classical scales used to measure the treatment effects, all patients will be examined using a functional magnetic resonance imaging (fMRI) before and after treatment to explore the cerebral effects of rTMS

DETAILED DESCRIPTION:
Repetitive Transcranial Magnetic Stimulation (rTMS) has been shown to be an effective therapeutic tool for the treatment of several neuropsychiatric disorders including major depression and hallucinations in schizophrenia but, to date, studies exploring the effects of rTMS in Obsessive Compulsive Disorder (OCD) have produce negative or conflicting results, especially those applying the stimulation to the prefrontal cortex as for the treatment of depression. However, a promising result has been obtained in a study in which the rTMS was applied to the Supplementary Motor Area (SMA), but in a small size and heterogeneous sample. The SMA has connections with areas of the brain, especially motor areas and subcortical-limbic circuitry, implicated in OCD.

In our study, 40 adult outpatients with OCD, who have been insufficiently responsive to at least two recognized drug treatments, will be randomly assigned to one of two treatment groups (active low frequency (1 Hz, 100% of the motor threshold) rTMS or sham-placebo) applied to the SMA daily for up to four weeks. An individual MRI-guided neuronavigation will be used to precisely define the target stimulation site in each patient. Rating scales for symptom change will be obtained at baseline, during the rTMS course, at the end of 4 weeks of treatment, and after a 2-month follow-up period. The main outcome measure will be the Yale-Brown Obsessive Compulsive scale, and secondary outcome measure will include the CGI scales, the LPO scale, the MOCI, and the SDS. Brain activity changes in fMRI before and after active/sham treatment will be compared between groups, with rest measures and provocation tasks.

ELIGIBILITY:
Inclusion Criteria:

* signed patient informed consent;
* primary obsessive compulsive disorder;
* current YBOCS score at least 15 with or without drug (or obsessive/compulsive subscores of at least 10);
* males/females 18-65yrs;
* treated with at least two adequate dose of SRI at least 8 weeks at some stage of illness;
* currently using adequate, stable dose of SSRI at least 8 weeks but not responding.

Exclusion Criteria:

* schizophrenia, other psychotic disorders, bipolar I, current major depressive disorder (MADRS>20), substance/alcohol dependence within last 6 months;
* severe axis II;
* significant suicide risk;
* metallic implant in cranium;
* severe/unstable medical conditions;
* ECT in the last month;
* pregnancy or breastfeeding ;
* history epilepsy; neurological disorder leading to increased intracranial pressure; severe cardiac disorder/intracardiac lines, pacemakers; Gilles de la Tourette syndrome;
* current structured psychotherapy;
* current drug treatment of bipolar disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (YBOCS) | week 1, 2, 3, 4, 5, 7, 9, 11, 13

SECONDARY OUTCOMES:
Clinical Global Impression - Severity (CGI-S) | week 1, 2, 3, 4, 5, 7, 9, 11, 13
- Clinical Global Impression - Improvement (CGI-I) | week 1, 2, 3, 4, 5, 7, 9, 11, 13
Global Assessment of Functioning (GAF) | week 5, 13
- Montgomery Asberg Depression Rating Scale (MADRS) | week 5, 13
Brief Anxiety Scale (BAS | week 5, 13
Sheehan Disability Scale (SDS) | , week 5, 13
Hospital Anxiety and Depression (HAD) scale | week 1, 2, 3, 4, 5, 7, 9, 11, 13
Maudsley Obsessional Inventory (MOCI) | week 5, 13
LPO scale | week 5, 13

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Pelissolo, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Pitie Salpetriere Hospital, Paris, France